CLINICAL TRIAL: NCT01789827
Title: Interleukin-2 Imaging as a Guide to Cancer Immunotherapy (Ipilimumab or Pembrolizumab) in Advanced Melanoma: A Pilot Study
Brief Title: Aldesleukin Imaging in Viewing Tumor Growth in Patients With Stage IV Melanoma Receiving Ipilimumab or Pembrolizumab Therapy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MC1274; NCI-2013-00297 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Mod12-003605-14; MC1274 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2013-02-08; First posted 2013-02-12 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-04

CONDITIONS: Stage IV Skin Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort I (scintigraphy prior to immunotherapy and 12 weeks) (Experimental): Patients undergo technetium Tc 99 hydrazinonicotinamide-tricine-linked interleukin-2 scintigraphy prior to receiving ipilimumab or pembrolizumab and at 12 weeks.
  Interventions: Other: Laboratory Biomarker Analysis; Procedure: Radionuclide Imaging; Biological: Technetium Tc 99 Hydrazinonicotinamide-Tricine-linked Interleukin-2
- Cohort II (scintograpy prior to immunotherapy, 3-4, 12 weeks) (Experimental): Patients undergo technetium Tc 99 hydrazinonicotinamide-tricine-linked interleukin-2 scintigraphy prior to receiving ipilimumab or pembrolizumab, at 3-4 weeks, and at 12 weeks.
  Interventions: Other: Laboratory Biomarker Analysis; Procedure: Radionuclide Imaging; Biological: Technetium Tc 99 Hydrazinonicotinamide-Tricine-linked Interleukin-2

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Radionuclide Imaging — Undergo technetium Tc 99 hydrazinonicotinamide-tricine-linked interleukin-2 scintigraphies
  Other Names: nuclear medicine scan; radioimaging; Radionuclide Scanning; Scan; SCINTIGRAPHY
Biological: Technetium Tc 99 Hydrazinonicotinamide-Tricine-linked Interleukin-2 — Undergo technetium Tc 99 hydrazinonicotinamide-tricine-linked interleukin-2 scintigraphies
  Other Names: 99mTc-HYNIC-IL2

SUMMARY:
This pilot clinical trial studies aldesleukin imaging in viewing tumor growth in patients with stage IV melanoma receiving ipilimumab or pembrolizumab therapy. Diagnostic procedures, such as single-photon emission computed tomography (SPECT), uses radioactive drugs and a scanner to make detailed pictures of areas inside the body and may be a less invasive way to check for stage IV melanoma. Radioactive drugs, such as technetium Tc 99 hydrazinonicotinamide-tricine-linked interleukin-2, carry radiation directly to cancer cells and may be able to differentiate between tumor growth due to inflammation versus tumor progression in patients with stage IV melanoma receiving therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Feasibility/biodistribution of 99mTc-HYNIC-IL2 (technetium Tc 99 hydrazinonicotinamide-tricine-linked interleukin 2) scintigraphy in patients with metastatic melanoma undergoing immunotherapy with either ipilimumab (commercial source) or pembrolizumab.

SECONDARY OBJECTIVES:

I. Correlation of tumor infiltrating lymphocyte (TIL) invasion (scintigraphy/histology) with tumor burden; and description of any clinical side effects associated with imaging.

TERTIARY OBJECTIVES:

I. Correlation of TIL invasion assessed by 99mTc-HYNIC-IL2 scintigraphy vs. histology (total and subsets of TIL), as well as screen for peripheral blood correlates.

OUTLINE: Patients are assigned to 1 of 2 groups. COHORT I: Patients undergo technetium Tc 99 hydrazinonicotinamide-tricine-linked interleukin-2 scintigraphy prior to receiving ipilimumab or pembrolizumab and at 12 weeks.

COHORT II: Patients undergo technetium Tc 99 hydrazinonicotinamide-tricine-linked interleukin-2 scintigraphy prior to receiving ipilimumab or pembrolizumab, at 3-4 weeks, and at 12 weeks.

After completion of study treatment, patients are followed up at 30-45 days.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic proof of stage IV melanoma (pathology report confirmation) with plans to initiate therapy with ipilimumab or pembrolizumab according to Food and Drug Administration (FDA) approved guidelines, with multiple lesions such that

  * Two of these lesions are in the same organ and at least one of these two lesions is measurable by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 using either intravenous (IV) contrast enhanced computed tomography (CT) or CT component of positron emission tomography (PET)/CT OR
  * Three of these lesions are in different organs and at least one of these 3 lesions is measurable by RECIST 1.1 using either IV contrast enhanced CT or CT component of PET/CT
* Patient eligible for and will be receiving ipilimumab or pembrolizumab as standard of care therapy
* Absolute neutrophil count (ANC) >= 1500 mL
* Hemoglobin (Hgb) > 10 g/dL
* Platelets (PLT) >= 50,000 mL
* Aspartate aminotransferase (AST) =< 3 x upper limit of normal (ULN)
* Alkaline phosphatase =< 3 x ULN; up to 5 x allowed for patients with liver metastases
* Ability to provide informed consent
* Willingness to return to Mayo Clinic Rochester for follow-up
* Life expectancy >= 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* For women of childbearing potential, a negative serum pregnancy test =< 7 days prior to registration
* Willingness to participate in mandatory imaging studies as well as provide mandatory blood samples for correlative research
* Tumor accessible for biopsy

Exclusion Criteria:

* Uncontrolled or current infection
* Known allergy to 99mTc-HYNIC-IL2 or components
* Any of the following prior therapies with interval since most recent treatment:

  * Chemotherapy =< 3 weeks prior to registration
  * Biologic therapy =< 3 weeks prior to registration
  * Radiation therapy =< 3 weeks prior to registration
* Failure to recover from side effects of prior chemotherapy or surgery
* Any of the following:

  * Pregnant women
  * Nursing women
  * Women of childbearing potential or their sexual partners who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-06-27 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who develop scintigraphy limiting toxicities (SLTs) | Up to 12 weeks
  SLTs include grade 2+ allergic reaction, grade 3+ anaphylaxis, grade 2+ injection site reaction, or grade 3+ non-hematologic toxicity (not attributed to immunotherapy treatment/progression or a co-morbid condition). A 95% binomial confidence interval of the proportion of patients who develop a grade 2+ allergic reaction, grade 3+ anaphylaxis, or grade 2+ injection site reaction will be constructed.

SECONDARY OUTCOMES:
Incidence of adverse events, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 30-45 days after study discontinuation
  The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns.
Target-to-background (T/B) ratio as determined by technetium Tc 99 hydrazinonicotinamide-tricine-linked interleukin-2 scintigraphy | Up to 12 weeks
  Spearman rank correlation coefficients will be used to examine the association between T/B ratio and the pre-treatment tumor biomarkers. Spearman rank correlation coefficients will be used to examine the association between changes in T/B ratio, changes in TIL percentages, and changes in peripheral blood concentrations of T, B, and NK cell subsets.
TIL invasion as determined by technetium Tc 99 hydrazinonicotinamide-tricine-linked interleukin-2 scintigraphy | Up to 12 weeks
  Relationship between TIL invasion, tumor burden, tumor based biomarkers, and peripheral blood biomarkers will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Svetomir Markovic, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States